CLINICAL TRIAL: NCT01757132
Title: Post-approval Study of VisionCare's Implantable Miniature Telescope (by Dr. Isaac Lipshitz) in Patients With Bilateral Severe to Profound Central Vision Impairment Assoc. With End-stage Age-related Macular Degeneration
Brief Title: Post-Approval Study of the Implantable Miniature Telescope
Acronym: PAS-01
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VisionCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PAS-01
Record Dates: First submitted 2012-11-13; First posted 2012-12-28 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: AMD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implantable Miniature Telescope (Other): Post approval study
  Interventions: Device: Implantable Miniature Telescope

INTERVENTIONS:
Device: Implantable Miniature Telescope — Device - Implantable Miniature Telescope

SUMMARY:
The objective of the PAS-01 study is to assess the safety of the intraocular as measured by the cumulative incidence of patients who within 5 years after implantation experience persistent vision-impairing corneal edema (corneal edema leading to persistent loss of best corrected distance visual acuity >2 lines from pre-surgery baseline level).

The study will test the null hypothesis that the percentage of patients who experience persistent vision-impairing corneal edema is >17% against the alternative that the percentage is <17%. The null hypothesis will be rejected if the upper bound of the two-sided 95% confidence integral for the observed percentage is <17%.

DETAILED DESCRIPTION:
ECD sub-study. At investigative sites participating in the ECD Sub-Group study, corneal endothelial cell density will be measured by non-contact specular microscopy in a subgroup of 150 patients enrolled in the IMT-PAS-01 in the eye schedule for and implanted with the intraocular telescope at study entry, 3 months, 12, months, 24 months, 36 months, 48 months and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* stable severe (BVDCA of 10/160 or poorer) to profound (BCDVA of 20/800 or better) vision impairment caused by bilateral central scotomas associated with end-stage age-related macular degeneration.
* 65 years of age or older
* retinal findings of geographic atrophy or disciform scar with foveal involvement
* visually significant cataract
* agree to undergo pre- and post-surgery training and assessment
* achieve at least a 5-letter improvement with external telescope
* have adequate peripheral vision in the eye not scheduled for surgery

Exclusion Criteria:

* Stargardt's macular dystrophy
* Anterior chamber depth < 3.0mm
* Presence of corneal guttate
* Do not meet minimum age and endothelial cell density requirements
* evidence of CNV or treatment of CNV within the past 6 months
* cognitive impairment that would interfere with ability to understand and complete Acceptance of Risk and Informed Decision Agreement or prevent proper training/rehabilitation
* previous intraocular or cornea surgery of any kind in operative eye, including any type of surgery for either refractive or therapeutic purposes or who have prior or expected ophthalmic related surgery within 30 days preceding intraocular telescope surgery
* history of steroid-responsive rise in intraocular pressure, uncontrolled glaucoma, or preoperative IOP >22 mm Hg while on maximum medication
* known sensitivity to post-operative medications
* history of eye rubbing or an ocular condition that predisposes eye rubbing
* myopia >6.0 D
* hyperopia >4.0D
* axial length <21mm
* narrow angle, i.e., <Schaffer grade 2
* cornea stromal or endothelian dystrophies, including guttate
* inflammatory ocular disease
* zonular weakness/instability of crystalline lens, or pseudoexfoliation
* diabetic retinopathy
* untreated retinal tears
* retinal vascular disease
* optic nerve disease
* history of retinal detachment
* intraocular tumor
* retinitis pigmentosa

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2010-08; Primary Completion 2023-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Long term safety study of implantable miniature telescope | 5 years after implantation
  Number of persistent vision impairing corneal edema adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Oliver D Schein, MD, Principal Investigator — Johns Hopkins University
Locations (16):
- United States (16):
  - Arizona Eye Center, Chandler, Arizona
  - Retinal Consultants of Arizona, LTD, Phoenix, Arizona
  - Barnet, Dulaney, Perkins Eye, Phoenix, Arizona
  - Retina-Vitreous Associates, Beverly Hills, California
  - Retina Consultants of Orange County, Fullerton, California
  - Loma Linda University Health Care, Loma Linda, California
  - University of California - Davis, Sacramento, California
  - Specialty Eye Care (Glaucoma Consultants of Colorado), Parker, Colorado
  - Retina Speciality Institute, Pensacola, Florida
  - Sarasota Retinal Institute, Sarasota, Florida
  - Emory Eye Center, Atlanta, Georgia
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Pepose Vision Institute, Chesterfield, Missouri
  - New York Eye & Ear, New York, New York
  - Fine, Hoffman & Packer, Eugene, Oregon
  - Valley Retina Institute, McAllen, Texas